CLINICAL TRIAL: NCT05972538
Title: Clinical Performance and Stability of Different Types of Implant Supported Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Asmaa Nabil Elboraey, Associate Professor, National Research Centre, Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 64312012023
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Complete Edentulism
Keywords: Implant stability; Pocket depth; Patient Satisfaction; Overdentures
MeSH Terms: conditions — Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: two groups.Group I received ball and socket retained mandibular implant overdenture while Group II received cement retained implant supported fixed bridges
Who Masked: Participant
Masking Description: participants don't know which treatment type they received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): patients received ball and socket retained mandibular implant overdentures restoring complete edentulous mandible.
  Interventions: Device: Osstell ( Osstell AB, Goteborg, Sweden).; Device: periodontal probe (Vivacare, TPS, Vivadent, Schaan, Lichtenstein; Other: questionnaire for patient satisfaction
- Group II (Experimental): patients received cement retained mandibular implant overdentures restoring complete edentulous mandible.
  Interventions: Device: Osstell ( Osstell AB, Goteborg, Sweden).; Device: periodontal probe (Vivacare, TPS, Vivadent, Schaan, Lichtenstein; Other: questionnaire for patient satisfaction

INTERVENTIONS:
Device: Osstell ( Osstell AB, Goteborg, Sweden). — Implant stability were assessed on 15, 30,60 and 90 days of prosthesis delivery
Device: periodontal probe (Vivacare, TPS, Vivadent, Schaan, Lichtenstein — Clinical evaluation included assessment of pocket depth, plaque index and bleeding on probing) around the implant abutments on 15, 30,60 and 90 days of prosthesis delivery
  Other Names: - Assessment of implants clinical performance
Other: questionnaire for patient satisfaction — A questionnaire was used to evaluate patient satisfaction on 90 days at the end of follow up period.

SUMMARY:
A Total number of 36 implants were installed in 6 patients having mandibular single denture.

The patients were divided into two groups according to the definitive prosthesis.

Group I received ball and socket retained mandibular implant overdenture while Group II received cement retained implant supported fixed bridges.

DETAILED DESCRIPTION:
Implant's stability, clinical performance (gingival index, pocket depth, plaque index and bleeding on probing) and patient's satisfaction were performed after 15, 30,60 and 90 days after prosthesis delivery

ELIGIBILITY:
Inclusion Criteria:

* highly co-operative
* non-smoker
* systemically free from any chronic diseases

Exclusion Criteria:

* immunocompromised patients
* patients having knife edge, flat or flabby ridge,
* patients having T. M. J disorders

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Assessment of change in implant stability | on the 15th, 30th, 60th and 90th days of overdenture insertion
  Assessment of implant stability by device ( Ostell device)
Assessment of change in implants clinical performance throughout the follow-up period. | on the 15th, 30th, 60th and 90th days of over denture insertion.
  Assessment of change in pocket depth, plaque index and bleeding on probing) around the implant abutments. by periodontal probe.

SECONDARY OUTCOMES:
Assessment of patient satisfaction | on the 90th day of prosthesis delivery
  A questionnaire was used to evaluate patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa N. Elboraey, Asso, Prof, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Dokki, Egypt